CLINICAL TRIAL: NCT04998175
Title: Multi-omics Research of Prognostic Factors of Ventriculoperitoneal Shunt for Idopathic Normal Pressure Hydrocephalus
Brief Title: Multi-omics Research of Idopathic Normal Pressure Hydrocephalus (iNPH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Westlake University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-796
Record Dates: First submitted 2021-06-21; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: Idiopathic Normal Pressure Hydrocephalus; Prognostic factor; Ventriculoperitoneal shunt; Cerebrospinal fluid; Proteomics
MeSH Terms: interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNPH cohort (Experimental): The patients diagnosed of iNPH.
  Interventions: Procedure: ventriculo-peritoneal shunt

INTERVENTIONS:
Procedure: ventriculo-peritoneal shunt — A ventriculoperitoneal shunt is a tube that drains excess cerebrospinal fluid into abdomen

SUMMARY:
The research is designed to study the prognostic factors of ventriculoperitoneal (VP) shunt for iNPH by multi-omics research

DETAILED DESCRIPTION:
Preoperative T1-MRI, functional MRI and diffusion MRI imaging data of iNPH patients were collected. The clinical assessment was performed before/after the lumbar puncture test and 6 months after VP shunt. Clinical assessment included Mini-mental State Examination (MMSE), gait scores, Kiefer score, and Modified Rankin Scale (mRS). The cerebrospinal fluid was collected by tap-test, and 6 months after surgery by puncturing in the VP device pump.

Methods- The primary methods used are:

1. The cerebrospinal fluid proteomic analysis of iNPH patients before and after VP shunt surgery.
2. The structral and functional MRI analysis of iNPH patients
3. The clinical assessment of MMSE, gait scores, Kiefer score, and mRS. Objective- To study the prognostic factors of VP shunt for iNPH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years;
* Diagnosis of iNPH based on clinical assessment
* Participant is able to give written informed consent

Exclusion Criteria:

* Combining AD and Parkinson's disease and other nervous system diseases
* Participant is not medically available for shunt surgery
* Secondary NPH

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Proteomic pattern of CSF in iNPH patients | Before surgery in lumbar CSF
  Comparing the proteomic pattern differences in CSF between iNPH patients and normal age-matched normal volunteers by the analysis of mass spectrometry. Also, the responsive and non-responsive iNPH patients proteomic pattern were analzed.
Proteomic pattern changes of CSF in iNPH patients after VP shunt | Change from Baseline (ventricular CSF) at 6 months after VP shunt
  Comparing the proteomic pattern differences in CSF of iNPH patients before surgery and after VP shunt by the analysis of mass spectrometry. Also, the responsive and non-responsive iNPH patients proteomic pattern were analzed.

SECONDARY OUTCOMES:
Gray Matter Density | Before surgery
  Using automatic cortical and subcortical segmentation from the 3-dimensional T1weighted images to measure gray matter density in iNPH patients before surgery compared with healthy individual group. Also, the responsive and non-responsive iNPH patients structral MRI were analzed.
Change in the resting state fMRI | Before surgery
  Change of BOLD singal intensity in the resting state fMRI in iNPH patients compared with normal healthy group. Also, the responsive and non-responsive iNPH patients functional MRI were analzed.
White matter abnormity | Beore surgery
  Franctional anisotropy, mean diffusivity and apparent diffusion coefficient were measured by diffusion MRI in region of interest of iNPH patients compared with normal healthy group. Also, the responsive and non-responsive iNPH patients diffusion MRI were analzed.
Kiefer score | Change from Baseline at 6 months after VP shunt
  A score for iNPH severity; range 0-26; higher indicates higher severity.
Mini mental state Examination | Change from Baseline at 6 months after VP shunt
  A score for cognitive ability; range 0-30; higher indicates higher severity.
Gait evaluation | Change from Baseline at 6 months after VP shunt
  10 meters walking test were evaluated of iNPH patients.
modified Rankin scale | Change from Baseline at 6 months after VP shunt
  A score for functional neurological status ; range 0-5; higher indicates higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Zhoule Zhu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The second affliated hospital of zhejiang university, Hangzhou, Zhejiang, China